CLINICAL TRIAL: NCT05183100
Title: Effects of Neurodynamics on Lower Extremity Spasticity - a Study in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: YM110045E
Record Dates: First submitted 2021-12-05; First posted 2022-01-10 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2021-10

CONDITIONS: Chronic Stroke; Stroke; Spasticity Post Stroke
Keywords: Neurodynamics; Calf muscle spasticity; Chronic stroke
MeSH Terms: conditions — Stroke | interventions — Supine Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (Neurodynamics Treatment) (Experimental): Neurodynamic treatment for about 13 minutes in supine position. It will be comprised of three stages, and the tensioner technique of the tibial nerve will be used.
  Interventions: Procedure: Tibial Nerve Neurodynamics
- Control Condition (Active Comparator): Lying in supine.
  Interventions: Procedure: Lying in supine

INTERVENTIONS:
Procedure: Tibial Nerve Neurodynamics — The patient will lie supine with the trunk and neck in neutral position. During the first stage, participants will receive passive straight leg raise of the affected side held for 20 seconds for 3 repetitions. In the second stage, hip adduction and internal rotation, ankle dorsiflexion, and ankle eversion are added in the straight leg raise position. Slow oscillations of the ankle movement for 1 minute will be applied, followed by holding the position for 20 seconds, for 3 repetitions. In the third stage, the head of the patient will be held in flexion with pillows while the same oscillation procedure as the second stage is performed. There will be a 2-minute rest between the stages.
  Other Names: Tibial Nerve Neural Mobilization
  Arms: Experimental Condition (Neurodynamics Treatment)
Procedure: Lying in supine — Lying in supine position for about 13 minutes.
  Arms: Control Condition

SUMMARY:
Post-stroke spasticity in the lower extremity affects balance and gait, leading to decreased mobility and functional independence. Therefore, effective intervention for reducing spasticity is crucial in stroke rehabilitation. Recently, neurodynamics, though originally designed for pain management in orthopedic patients, has also been applied for treating spasticity in patients with neurological disorders. However, previous studies focused mainly on treating the upper extremity spasticity, but not on lower extremity spasticity, and not on possible neurophysiological changes. The present study aims to investigate the immediate effects of neurodynamics in reducing lower limb spasticity and neurophysiological changes in people with chronic stroke.

DETAILED DESCRIPTION:
Sample size calculation: There was no reference for the effect size of neurodymanics on reducing lower extremity spasticity, and the effect size of neurodynamics treatment for improving knee range of motion was between 0.89 to 2.55. We set the effect size of 0.6 (moderate effect size) with an alpha level of 5%, power at 80%, and a paired t-test model to calculate the sample size.

Statistical analysis: Paired t-test will be used for within condition (experimental or control condition) comparisons. The change values between pre and post in each condition will be calculated and compared by paired t-test for between condition comparisons. The significance is set at p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first-ever stroke with unilateral lesion for more than 6 months
* demonstrating calf muscle spasticity as indicated by modified Ashworth scale equal to or greater than 1
* with passive ROM of ankle dorsiflexion at least to neutral position (defined as 0°)
* ability to walk at least 10m independently without a walking device or ankle-foot orthosis (AFO)
* sufficient cognition (mini-mental state examination, MMSE score of 24 or higher)

Exclusion Criteria:

* contraindications to nerve conduction tests
* other orthopedic and neurological disorders interfering participating in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Change in Spasticity: Clinical measurement | Before intervention and immediately after intervention
  The modified Ashworth scale (MAS) will be used, which is a 6-point scale commonly used to assess muscle spasticity in clinical settings.
Change in Spasticity: Neurophysiological measurement | Before intervention and immediately after intervention
  The H-reflex will be recorded by placing a disposable surface electrode on the muscle belly of the gastrocnemius after a stimulation of the tibial nerve just proximal to the electrode.

SECONDARY OUTCOMES:
Change in Gait Performance | Before intervention and immediately after intervention
  Gait performance will be measured by using the GAITRite system (CIR system, Inc., Havertown, Pennsylvania). Participants will be instructed to walk along the walkway at their comfortable speed. Gait velocity, cadence, and step length of the affected and unaffected limbs, and spatial and temporal asymmetry ratios are calculated.
Change in Lower Extremity Motor Control | Before intervention and immediately after intervention
  Motor control of the lower extremity will be assessed by the motor section of the Fugl-Meyer Assessment (FMA). Higher scores represent better motor control, with a total score of 34.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez Lopez L, Torres JR, Rubio AO, Torres Sanchez I, Cabrera Martos I, Valenza MC. Effects of neurodynamic treatment on hamstrings flexibility: A systematic review and meta-analysis. Phys Ther Sport. 2019 Nov;40:244-250. doi: 10.1016/j.ptsp.2019.10.005. Epub 2019 Oct 15. PMID 31655484
- [Background] Cha HK, Cho HS, Choi JD. Effects of the nerve mobilization technique on lower limb function in patients with poststroke hemiparesis. J Phys Ther Sci. 2014 Jul;26(7):981-3. doi: 10.1589/jpts.26.981. Epub 2014 Jul 30. PMID 25140078
- [Background] Datta Gupta A, Visvanathan R, Cameron I, Koblar SA, Howell S, Wilson D. Efficacy of botulinum toxin in modifying spasticity to improve walking and quality of life in post-stroke lower limb spasticity - a randomized double-blind placebo controlled study. BMC Neurol. 2019 May 11;19(1):96. doi: 10.1186/s12883-019-1325-3. PMID 31078139